CLINICAL TRIAL: NCT02548871
Title: Evaluation of the Teen Outreach Program in Chicago Public Schools: Replication of an Evidence-Based Teen Pregnancy Prevention Program
Brief Title: Evaluation of the Teen Outreach Program in Chicago Public Schools
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Chapin Hall at the University of Chicago (Other)
Collaborators: Chicago Public Schools (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Prevention
Other Study IDs: TP1AH000066
Record Dates: First submitted 2015-09-10; First posted 2015-09-14 (Estimated); Last update posted 2015-09-14 (Estimated); Status verified 2015-09

CONDITIONS: Sexual Behavior
MeSH Terms: conditions — Sexual Behavior

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- Teen Outreach Program (Experimental): Teen Outreach Program
  Interventions: Behavioral: Teen Outreach Program
- Comparison (No Intervention): Business as usual

INTERVENTIONS:
Behavioral: Teen Outreach Program — TOP® is a positive youth development and service learning program for youth ages 12 to 17, and its Changing Scenes curriculum is separated into age appropriate levels. The program uses an approach that involves a caring adult, positive self-efficacy, future planning and goal setting and life management skills to to reduce risky sexual behavior and improve school outcomes. TOP® is designed to be delivered in weekly sessions over 9 months and includes community service learning.
  Arms: Teen Outreach Program

SUMMARY:
The purpose of this study was to determine the impact of TOP® on sexual health behavior.

DETAILED DESCRIPTION:
The cluster-randomized study was conducted in 9th grade classrooms in Chicago Public Schools (CPS) with equal number of schools randomized to intervention and comparison groups for two cohort years. Students were administered a scannable paper survey at three time points: baseline, post-program and 1-year post program. The primary impact analysis used an intent-to-treat approach. Implementation of TOP® was assessed by conducting classroom observations. TOP® was delivered in a variety of classroom settings over the school year by facilitators from CPS and partner organizations.

ELIGIBILITY:
Inclusion Criteria:

* First-time 9th grade student
* Passive parental consent and student assent

Exclusion Criteria:

* Inability to complete survey in languages provided

Ages: 12 Years to 17 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Child
Enrollment: 12253 (Actual)
Dates: Start 2010-09; Primary Completion 2014-06 (Actual); Study Completion 2015-08 (Actual)

PRIMARY OUTCOMES:
Sex without a condom in the last 90 days | 9 months after baseline
  Dichotomous indicator from self-report survey

SECONDARY OUTCOMES:
Sex in the last 90 days | 9 months after baseline
  Dichotomous indicator from self-report survey
Sex without a condom in the last 90 days, by race/ethnicity | 9 months after baseline
  Dichotomous indicator from self-report survey
Sex without a condom in the last 90 days | 21 months after baseline
  Dichotomous indicator from self-report survey

REFERENCES:
- [Background] Seshadri R, Smithgall C, Goerge R, Ippolito J, Dasgupta D, Wiegand E, Guiltinan S, Wood M. (2015) Evaluation of the Teen Outreach Program: Findings from the Replication of an Evidence-Based Teen Pregnancy Prevention Program. Chicago, IL: Chapin Hall at the University of Chicago